CLINICAL TRIAL: NCT05418205
Title: Strengthening and Relieving the Burden on Families With Children in Need of Care Through Family Health Partners [Familien-Gesundheits-Partner; FGP] in Regional Network Structures
Brief Title: Family Health Partners in Regional Network Structures
Acronym: NEST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Federal Joint Committee (Other Government); aQua-Institut GmbH, Germany (Unknown); Leibniz-Institut für Resilienzforschung, Germany (Unknown); nestwärme gGmbH, Germany (Unknown); Kindernetzwerk e.V., Germany (Unknown); ism gGmbH, Germany (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 01VSF20004
Record Dates: First submitted 2022-03-01; First posted 2022-06-14 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Disabled or Chronically Ill Children in Need of Care
Keywords: children in need of care; family caregivers; Family Health Partner; non-medical care; regional networking

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (IG) (Experimental): Families with FGP support (families with disabled and/or chronically children under 18 in the greater area of Mainz, Saarbrucken and Munich (Germany)
  Interventions: Other: Families with FGP support
- Control Group (CG) (No Intervention): Families without FGP support (standard care) under the same conditions

INTERVENTIONS:
Other: Families with FGP support — Non-randomized controlled trial with four points of measurement ( in 18 months)
  Arms: Intervention Group (IG)

SUMMARY:
Families with children with severe health problems are exposed to particular emotional, social, economic and time burdens. These result in further risks, which often lead to poor living and care situations for the families concerned. This is attributed, among other, to legal regulations that do not do justice to the respective individual life situations and the lack of competent information and counselling services. The overarching objective of the NEST project is to evaluate the effectiveness of a professional support facility for families with children in need of care that operates across sectors and service providers. The network support by so-called Family Health Partners [Familien-Gesundheits-Partner; FGP] aims to provide assistance and need-based individual care for all members in families with children in need of care. The medium-term goal of FGP support is to develop the family as a self-help system, i.e. as a self-competent, independently acting primary resource for the care and support of their children in need of care.

DETAILED DESCRIPTION:
The project starts facing the problem that families with children with severe health problems are exposed to strong emotional, social, economic and temporal burdens. This results in further health, social and economic risks, which often lead to poor living and care situations for the families concerned. This is attributed, among other things, to legal regulations that do not do justice to the respective individual life situations and the lack of competent advice and contact points. The overarching objective of the NEST project is the evaluation of an innovative support service that addresses the problem. The network support by so-called Family Health Partners [Familien-Gesundheits-Partner; FGP] aims to provide needs-based, individual care for all members in families with children in need of care, i.e. the best possible physical, psychological and participation-oriented care for children in need of care, thus relieving the relatives who spend much time for care and assistance of their child/children. The intervention to be evaluated here with regard to its effectiveness and to be analyzed with regard to its impact factors (processes and structures) was summarized in the term of FGP. This personalized function, which is anchored in the network, aims to provide "holistic" support for families with children in need of care. This means that the needs of the families are determined individually and initially independent of sectoral or service provider specific offers (structured assessment). The needs of families not only relate to medical, nursing or therapeutic care, but also to assistance regarding social law, economic and bureaucratic advice as well as social, psychosocial and emotional needs and social participation. Based on the identified need for support, affected families are individually accompanied by FGP over a certain period of time (in the project context: a maximum of 18 months). The medium-term goal of FGP support is to strengthen or maintain the family as a self-help system, i.e. self-efficient, independently acting primary resource for the care and support of their children (preventive).

ELIGIBILITY:
Inclusion Criteria:

* parents and other guardians with at least one disabled and/or chronically ill child under 18 years in western and southern Germany
* all genders and ethnicities will be included in the study

Exclusion Criteria:

* caregivers for children in need of care according to § 37 of Germany's Social Security Code V level of care = 1 (i.e. minor impairments of independence or abilities)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Family quality of life | 18 months
  Name of the measurement and measurement tools can be seen below (outcome measures 2-9). Unit of measure are both measures of central tendency and measures of variability.
Parents' mental and physical health | 18 months
  General Health Questionnaire-28 - GHQ-28
Well-being | 18 months
  WHO-Five Well-being Index - WHO-5
Stress experience | 18 months
  Perceived Stress Scale - PSS-4
Family burden due to illness of the child | 18 months
  Impact-on-Family Scale - IOFS-20
Family cohesion | 18 months
  Resilience Scale for Adults - RSA
Resilience | 18 months
  Brief Resilience Scale - BRS
Individual stressor exposure | 18 months
  Mainz Inventory of Microstressors - MIMIS
Life events | 18 months
  Life History Calendar - LHC

SECONDARY OUTCOMES:
Resilience factors and associated measures | 18 months
  Name of the measurement and measurement tools can be seen below (outcome measures 11-14). Unit of measure are both measures of central tendency and measures of variability.
Optimism / positive thinking | 18 months
  Scale Optimism-Pessimism-2 - SOP-2
Locus of control | 18 months
  Internal and External Locus of Control Scale-4 - IE-4
Self-efficacy | 18 months
  General Self-efficacy Short Scale - ASKU-3
Social support | 18 months
  Oslo Social Support Scale - OSSS-3
Access to care | 18 months
  Operationalization see below (outcome measures 16-18).
Satisfaction with health care | 18 months
  Self-developed questionnaire with 13 items
Use of support services | 18 months
  Self-developed questionnaire with 21 items
Satisfaction with health coordination | 12 months
  Case Management questionnaire with 11 items

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Willms, PhD, Study Director — aQua-Institut GmbH, Germany
Locations (2):
- Germany (2):
  - Kindernetzwerk e.V., Mainaschaff
  - Nestwärme gGmbH, Trier

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Broll J, Schafer SK, Ludecke D, Nickel S, Lieb K, Helmreich I. Effects of micro- and macro-stressors and resilience factors on the mental health of parents caring for chronically ill and disabled children and adolescents. BMC Nurs. 2025 May 2;24(1):489. doi: 10.1186/s12912-025-03125-6. PMID 40316988
- [Derived] Nickel S, Helmreich I, Broll J, Ludecke D. Family health partners in regional network structures (NEST): A non-randomized controlled trial among parents of chronically ill and disabled children. PLoS One. 2023 Jul 17;18(7):e0288435. doi: 10.1371/journal.pone.0288435. eCollection 2023. PMID 37459306
- See also: Research project N.E.S.T. — https://www.forschungsprojekt-nest.de